CLINICAL TRIAL: NCT02549443
Title: The Anabolic Effect Of Perioperative Nutrition With Insulin In Patients Undergoing CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Roupen Hatzakorzian, MD, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-383-SDR
Record Dates: First submitted 2015-06-22; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Artery Disease
Keywords: Catabolic response; Amino Acids; Insulin
MeSH Terms: conditions — Coronary Artery Disease; Insulin Resistance | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Insulin (Active Comparator): hyperinsulinemic-normoglycemic clamp: an insulin infusion of 5 mU.kg-1.min-1 and a variable continuous infusion of glucose (dextrose 20%) to maintain the blood glucose between 4.0 and 6.0 mmol/L.
  Interventions: Dietary Supplement: Amino acids
- Insulin and amino acids (Active Comparator): hyperinsulinemic-normoglycemic clamp: an insulin infusion of 5 mU.kg-1.min-1 and a variable continuous infusion of glucose (dextrose 20%) to maintain the blood glucose between 4.0 and 6.0 mmol/L.
  Amino Acids (AA) in amounts to preserve normal AA
  Interventions: Dietary Supplement: Amino acids
- Insulin and hyperaminoacidemia (Active Comparator): hyperinsulinemic-normoglycemic clamp: an insulin infusion of 5 mU.kg-1.min-1 and a variable continuous infusion of glucose (dextrose 20%) to maintain the blood glucose between 4.0 and 6.0 mmol/L.
  AA in amounts to increase AA plasma concentrations to supra-normal levels (hyperaminoacidemia)
  Interventions: Dietary Supplement: Amino acids

INTERVENTIONS:
Dietary Supplement: Amino acids — AA (Travasol Baxter, Deerfield IL) during and after surgery in an amount equivalent to 20% and 35% of the patient's energy expenditure (EE)

SUMMARY:
This study evaluates whether providing a nutritional intervention in the form of insulin, sugar and protein during and after open-heart surgery will increase the body's protein stores and maintain a normal level of blood sugar. The primary outcome will be Whole body protein balance which will be assessed by isotope tracer kinetics. Protein balance will be calculated as protein synthesis minus protein breakdown with positive values indicating anabolism and negative values catabolism. The preoperative measurements will be performed on the morning before the operation. Postoperative studies will be conducted two hours after surgery in the intensive care unit. Patients will be followed for 12 hours after surgery.

DETAILED DESCRIPTION:
Open heart surgery is associated with a catabolic response which is characterized by hyperglycemia and whole body protein loss. Results of a previous study demonstrated that a reduction in whole-body protein breakdown and synthesis in patients receiving insulin and isocaloric amounts of glucose (hyperinsulinemic-normoglycemic clamp, HNC) after coronary artery bypass graft (CABG) surgery. Because protein oxidation did not change and the circulating concentrations of amino acids decreased (hypoaminoacidemia) in the presence of insulin therapy whole-body protein balance remained negative, ie patients were still catabolic. The investigators hypothesize that this lack of anabolic effect is due to the absence of anabolic substrate supply (amino acids). The primary objective of this study is to test the hypothesis that insulin administered as part of a hyperinsulinemic-normoglycemic clamp during and immediately after CABG:

1. Will induce whole-body positive protein balance if supplemented with intravenous amino acids (AA) in amounts to preserve normal AA plasma concentrations (isoaminoacidemia), and
2. Will further enhance whole-body protein balance if combined with the infusion of AA in amounts to increase AA plasma concentrations to supra-normal levels (hyperaminoacidemia) The primary outcome, whole body protein balance, will be measured 2 hours after surgery in the intensive care unit. Secondary objectives include (1) measure hepatic albumin synthesis and (2) assess changes in the metabolic-endocrine milieu.

Methods: 30 patients scheduled for elective CABG surgery requiring cardiopulmonary bypass will be enrolled. Consenting patients will be divided randomly into 3 groups. Patients in group 1 will receive HNC from the beginning of surgery until the end of the eight-hour study period after surgery. No amino acids will be given. Patients in group 2 will receive HNC and AA (Travasol Baxter, Deerfield IL) during and after surgery in an amount equivalent to 20% of the patient's energy expenditure (EE) as measured before surgery to maintain isoaminoacidemia. Patients in group 3 will receive HNC and Travasol iduring and after surgery in an amount equivalent to 35% of the patient's EE to promote hyperaminoacidemia. HNC will consist of an insulin infusion of 5 mU/kg/min coupled with a variable infusion of glucose (dextrose 20%) to maintain normoglycemia (4-6 mmol/L). Whole body protein balance will be assessed by L-[1-13C]leucine tracer kinetics. Protein balance will be calculated as protein synthesis minus leucine rate of appearance (Ra) with positive values indicating anabolism and negative values catabolism. Whole body glucose metabolism will be assessed by stable isotope tracers [6,6-2H2]glucose. Hepatic albumin synthesis will be determined by using primed continuous infusion of L-[2H5]phenylalanine. The preoperative measurements will be performed on the morning before the operation. Postoperative studies will be conducted 2 hours after surgery in the intensive care unit. Patients will be followed for 12 hours after surgery. Whole body leucine kinetics between the two groups will be analyzed using ANOVA for repeated measurements. Statistical significance will be set as P<0.05. All p-values will be presented are 2-tailed.

Tracer kinetics:

Whole body leucine and glucose metabolism measurements were made under postabsorptive conditions on the day before surgery and, postoperatively, in the intensive care unit. Plasma kinetics of glucose and leucine, i.e. the glucose and leucine rate of appearance (Ra), leucine oxidation and non-oxidative leucine disposal, were determined by a primed constant infusion of tracer quantities of L-[1-13C]leucine and [6,6-2H2]glucose. Blood and expired air samples were collected, before the infusion, to analyze baseline enrichments. Priming doses of NaH13CO3 (1 µmol/kg, po), L-[1-13C]leucine (4 µmol/kg, iv) and [6,6-2H2]glucose (22 µmol/kg, iv), were administered followed by the infusion of L-[1-13C]leucine (0.06 µmol.kg-1.min-1) and [6,6-2H2]glucose (0.44 µmol.kg-1.min-1). For the determination of 13CO2 isotope enrichments four expired breath samples were taken after 150, 160, 170 and 180 minutes of isotope infusion.

Whole body leucine and glucose kinetics were calculated by the conventional isotope dilution technique using a two-pool random model during steady state conditions. At isotopic steady state the Ra of unlabeled substrate in plasma is derived from the plasma isotope enrichment, expressed as MPE, according to the following equation: Ra = I.(MPEinf/MPEpl - 1), where I is the infusion rate of the tracer, MPEinf is the enrichment of the tracer in the infusate and MPEpl is the tracer enrichment in plasma. The final MPE values represent the mean of all the MPE measurements during each isotopic plateau. Isotopic steady state conditions were regarded as valid when the CV of the MPE values at isotopic plateau was <5%.

At isotopic steady state leucine flux (Q) is quantified by the following formula: Q = S+O = B+I, where S is the rate of synthesis of protein from leucine, O is the rate of oxidation, B is protein breakdown and I is the dietary intake. Furthermore Q is equal to Ra (Ra = B+I) and the rate of disappearance (Rd; Rd = S+O). When tracer studies are done in fasting states, leucine flux equals B. The rate of protein synthesis is calculated by subtracting leucine oxidation from leucine flux (S = Q-O). Protein balance is calculated as protein synthesis minus leucine Ra with positive values indicating anabolism and negative values catabolism. Plasma [1-13C]α-KIC is used to calculate the flux and oxidation of leucine. The α-KIC is formed intracellularly from leucine and is released into the systemic circulation. It reflects the intracellular precursor pool enrichment more accurately than plasma leucine itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective CABG

Exclusion Criteria:

* Severe malnutrition (weight loss >20% in preceeding 3 months, low albumin level <35 g/L and body mass index <20 kg/m2), obesity (body mass index >35 kg/m2), chronic liver disease (cirrhosis, documented chronic viral hepatitis and abnormal liver function tests), left ventricular ejection fraction <30%, active cancer, dialysis, <18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Whole body protein balance which will be assessed by isotope tracer kinetics. | preoperative (morning before the operation), two hours after surgery in the intensive care unit
  Protein balance will be calculated as protein synthesis minus protein breakdown with positive values indicating anabolism and negative values catabolism. Patients will be followed for 12 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Roupen Hatzakorzian, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Omiya K, Sato H, Sato T, Wykes L, Hong M, Hatzakorzian R, Kristof AS, Schricker T. Albumin and fibrinogen kinetics in sepsis: a prospective observational study. Crit Care. 2021 Dec 17;25(1):436. doi: 10.1186/s13054-021-03860-7. PMID 34920728
- [Derived] Codere-Maruyama T, Schricker T, Shum-Tim D, Wykes L, Nitschmann E, Guichon C, Kristof AS, Hatzakorzian R. Hyperinsulinemic-normoglycemic clamp administered together with amino acids induces anabolism after cardiac surgery. Am J Physiol Regul Integr Comp Physiol. 2016 Dec 1;311(6):R1085-R1092. doi: 10.1152/ajpregu.00334.2016. Epub 2016 Oct 5. PMID 27707724